CLINICAL TRIAL: NCT02169245
Title: Relative Effects of Chronic Consumption of Egg Protein at Breakfast With and Without Fiber on Brain Neural Activation, Appetite, Glycemic and Lipemic Control and Self-selected Energy Intake
Brief Title: Effects of Protein and Fiber at Breakfast on Appetite, Blood Sugar, and Cholesterol
Acronym: PFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Professor, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1208012603
Record Dates: First submitted 2014-03-20; First posted 2014-06-23 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Brain Activity; Appetite; Ingestive Behavior; Glucose Control; Cholesterol
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Average Protein and Fiber at Breakfast (Experimental): Dietary control of protein and fiber intake at breakfast. Participants will eat a 400 kcal breakfast with an average amount of protein and fiber for this age group for 2 weeks.
  Interventions: Other: Dietary control of protein and fiber intake at breakfast
- Average Protein and High Fiber at Breakfast (Experimental): Dietary control of protein and fiber intake at breakfast. Participants will eat a 400 kcal breakfast with an average amount of protein and higher than average amount of fiber for this age group for 2 weeks.
  Interventions: Other: Dietary control of protein and fiber intake at breakfast
- High Protein and Average Fiber at Breakfast (Experimental): Dietary control of protein and fiber intake at breakfast. Participants will eat a 400 kcal breakfast with an average amount of fiber and higher than average amount of protein for this age group for 2 weeks.
  Interventions: Other: Dietary control of protein and fiber intake at breakfast
- Higher Protein and Fiber at Breakfast (Experimental): Dietary control of protein and fiber intake at breakfast. Participants will eat a 400 kcal breakfast with a higher than average amount of protein and fiber for this age group for 2 weeks.
  Interventions: Other: Dietary control of protein and fiber intake at breakfast

INTERVENTIONS:
Other: Dietary control of protein and fiber intake at breakfast — Participants will be provided breakfast meals for 4, 2 week long interventions. The intervention arms are 1) average protein and fiber, 2) average protein and high fiber, 3) high protein and average fiber, and 4) high protein and fiber.

SUMMARY:
The objectives of the research are to assess the effects of increased protein and fiber intake at breakfast on neural activation in brain regions associated with appetitive drive and reward-driven eating, measures of subjective appetite, and ingestive behavior in overweight adults. Additional outcomes of interest include the effects of the breakfast intervention on blood sugar and cholesterol profiles.

DETAILED DESCRIPTION:
The objectives of the research are to assess the effects of increased protein and fiber intake at breakfast on neural activation in brain regions associated with appetitive drive and reward-driven eating, measures of subjective appetite, and ingestive behavior in overweight adults. Additional outcomes of interest include the effects of the breakfast intervention on 24-hour glucose profile as well as fasting and postprandial glycemic and lipemic regulation. The investigators will test the effects of consuming breakfasts with normal protein/normal fiber (NPNF), normal protein/high fiber (NPHF), high protein/normal fiber (HPNF), and high protein/high fiber (HPHF) for two weeks in a randomized cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 21 - 45 years
* BMI 25-29.9 kg/m2

Exclusion Criteria:

* Irregular menstrual cycles
* current smoker
* medications or supplements that affect appetite
* pregnant or lactating
* not weight stable
* acutely ill
* diabetic
* claustrophobic
* any implantation unsafe in magnetic resonance imaging (MRI) environment

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Brain activation measured with functional magnetic resonance imaging and its association with measures subjective of appetite, self-selected daily energy intake, and energy intake at an ad libitum lunch. | 16 weeks
  Aim 1: Assess the effects of a higher than normal protein and fiber intake at breakfast on neural activation of brain regions associated with appetitive drive and reward-driven eating, measures subjective of appetite, self-selected daily energy intake, and energy intake at an ad libitum lunch.

SECONDARY OUTCOMES:
24-hour blood glucose profile | 16 Weeks
  Aim 2: Assess the effects of higher than normal protein and fiber intake at breakfast on 24-hour glucose profile using a continuous glucose monitoring system.
Fasting and postprandial blood glucose, insulin, and lipid concentrations | 16 Weeks
  Aim 3: Assess the effects of higher than normal protein and fiber intake at breakfast on fasting and postprandial glycemic and lipemic regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University Dept of Nutrition Science
Locations (2):
- United States (2):
  - InnerVision West/Purdue MRI Facility, West Lafayete, Indiana
  - Purdue University, West Lafayette, Indiana